CLINICAL TRIAL: NCT01909622
Title: A Randomized Trial of Milk Fortified With Vitamin D in Colombia
Brief Title: Trial of Vitamin D Fortified Milk
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Eduardo Villamor, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VDFORT
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: 25-hydroxyvitamin D Serum Concentrations
Keywords: Vitamin D; Milk fortification; Children; Colombia
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Vitamin D-fortified milk (Experimental): Skim milk fortified with 600 IU vitamin D3 / 250 mL
  Interventions: Dietary Supplement: Vitamin D
- Vitamin D-unfortified milk (Active Comparator): Unfortified skim milk
  Interventions: Dietary Supplement: No vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D
  Arms: Vitamin D-fortified milk
Dietary Supplement: No vitamin D
  Arms: Vitamin D-unfortified milk

SUMMARY:
Prevalence of VDD is high worldwide, even in sunbathed equatorial regions where it had not been suspected before. The most cost-effective method for reducing population-wide VDD is through fortification of commonly consumed foods. Nevertheless, the efficacy of fortification varies by dose, duration, and population characteristics; and it is currently unknown whether it could be an efficacious public health intervention to curb the VDD epidemic among children living in tropical areas. We propose to conduct a randomized, controlled, double blind trial to assess the effect of vitamin D3 fortification of milk on serum 25-hydroxyvitamin D concentrations in school-age children and their mothers in Bogotá, Colombia. Eighty families with a child participating in an ongoing cohort study will be randomized to receive one liter per day of either skim milk fortified with 600 IU vitamin D3 per 250mL or unfortified skim milk for a six-week period. Caregivers will be instructed to give the index child two cups of milk per day and to distribute the remaining milk to the rest of the family. We will measure serum 25(OH)D concentrations of the children and mothers at baseline and at the end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 144 and 174 completed months by the time of enrollment.
2. Intention to stay in the city for the next six weeks.
3. Children living with their biological mothers.
4. Families own a refrigerator.

Exclusion Criteria:

1. History of illness involving calcium or bone metabolism, including stones of the urinary tract.
2. Currently taking vitamin D supplements as treatment of any disease.
3. Receiving immunosuppressive therapy (oral corticosteroids, chemotherapy) during the previous year.
4. Known history of lactose intolerance or other contra-indications or aversion to milk intake.
5. Known hypercalcemia.

Ages: 144 Months to 174 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of 25-OH vitamin D | up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Mora, MSc, RD, Study Director — FINUSAD - Foundation for Research in Nutrition and Health; Henry Oliveros, MD, MSc, Study Director — University of La Sabana; Eduardo Villamor, MD, DrPH, Principal Investigator — University of Michigan
Locations (2):
- Colombia (2):
  - FINUSAD - Foundation for Research in Nutrition and Health, Bogotá
  - University of La Sabana, Chía